CLINICAL TRIAL: NCT05242731
Title: MonSter Study, Telemonitoring and Connected Care Applied to Multiple Sclerose
Brief Title: Telemonitoring and Connected Care Applied to Multiple Sclerose
Acronym: MonSter
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Isala (Other)
Responsible Party: Principal Investigator, Marlies Hoving, Dr, Isala
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MonSter75251
Record Dates: First submitted 2022-01-23; First posted 2022-02-16 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: Single center, randomized control, non inferiority trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Active Comparator): Studygroup: Working with MSmonitor and video calling. Complete research questionnaires every 3 months in the Case Report Form, Researchmanager.
  Interventions: Device: MSmonitor, a self-management/education program with e-health interventions; Device: Video calling program "Better-close"; Device: Researchmanager program
- Controlgroup (Active Comparator): Became care as usual (CAU), not working with MSmonitor or video calling. Complete research questionnaires every 3 months in the Case Report Form, researchmanager.
  Interventions: Device: Researchmanager program

INTERVENTIONS:
Device: MSmonitor, a self-management/education program with e-health interventions — A self-management/education program with e-health interventions
  Arms: Study group
Device: Video calling program "Better-close" — Video calling program.
  Arms: Study group
Device: Researchmanager program — Case Report Form, Datamanagement program

SUMMARY:
The investigators designed a new care concept based on a multi-modal version of the MSmonitor program, the 'MSmonitor-Plus and Video Calling Care' (MPVC). MPVC combines the self-management and education program MSmonitor with video consultations by using specific questionnaires designed for high-frequency/intensive self-assessments of MS patients.

'The overall objective of this study is to assess the feasibility and (cost)-effectiveness of MPVC compared to Care as Usual (CAU).

An RCT with two parallel groups will be conducted to compare the MPVC with a CAU in MS patients and their caregivers.

In this study, 208 MS patients will be included with follow-up measurements for two years (at baseline and every three months).

After randomization, 104 patients will be assigned to MPVC and 104 patients to CAU.

The study will consist of three parts: 1) a clinical effectiveness study, 2) a cost-effectiveness study, and 3) process evaluation.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is the most common neurological disorder (1:500-1000) in young adults. It has a profound impact on all aspects of human functioning.

The clinical picture is comprehensive fatigue and often cognitive problems that negatively influenced the quality of life, but also the consultations in the hospital.

MS is not curable. In recent years new treatments have become available. These are more effective (can slow down or even stop MS) but also have more side effects and are more expensive. Careful monitoring based on effectiveness and side effects is therefore important. The result is a high frequency of hospital visits and a great burden on the patient. This great burden is expressed in an increase in the fatigue and cognitive problems that are already present, so the consultation in the hospital provides less information and is less efficient than desired.

Research has also shown, for example, that the complaints that MS patients discuss are mainly from the last 2 weeks. Previous complaints thus remain out of the picture

The aim is to optimize care for MS patients and to improve their quality of life. The costs will also be considered. The telemonitoring will be done by MSmonitor-Plus program with video calling care (MPVC). The MS patients fill in specific questionnaires every 3 months in the MSmonitor Plus. The healthcare professionals (HCP) can view the answers remotely and coordinate the right care. If the telemonitoring shows that the patient is doing well, it can be decided that the patient does not have to come to the hospital for a check-up.

By actively involving MS patients in the MSMonitor-Plus by filling in these questionnaires every 3 months, the HCP get a better picture of the complaints.

All MS patients actively receiving treatment within Isala are eligible for this study. There is randomization in which telemonitoring is compared with standard treatment. One group, the control group (CG) (104) continues care as usual (CAU), the other group, the intervention group (IG) (104) receives MSMonitor Plus and video calling care (MPVC).

During the research, both groups fill in research questionnaires every 3 to 6 months in an electronic case report form (Research Manager). These questionnaires are about general health, MS, health care consumption, autonomy, and quality of life are compared afterward.

A cost-effectiveness analysis will be made of both groups. The study will last a total of 2 years for the participating patients. Previous studies have been done with MSM, but not for a long period.

ELIGIBILITY:
Inclusion Criteria:

The participant is an MS patient who is being treated within the Isala. Is 18 years of age or older Has digital skills

The caregiver is the caregiver of an MS patient Is older than 18 years

Exclusion Criteria:

The patient does not master the Dutch language. The patient has insufficient computer skills. Disabled adults are excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Because there are more women with MS than men (70% female - 30% male)
Enrollment: 208 (Estimated)
Dates: Start 2021-04-29 (Actual); Primary Completion 2024-04-29 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint is Multiple Sclerose Quality of Life (MSQuol54) | 2 years
  The primary endpoint (MSQoL-54) at which the value of telemonitoring is determined is t=2 years.The 2 composite summary scores are the MSQOL-54 Physical Health Composite Score and the MSQOL-54 Mental Health Composite Score, The highest range is 100, de lowest 0. The lower the outcome (0) the better the quality of life. The higher the outcome (100), the worse the quality of life.

SECONDARY OUTCOMES:
Impact on participation and autonomy (IPA) | 2 years
  An secondary outcome measure is the autonomy of the MS patient.
Work together on health (PIH) | 2 years
  Receiving care that suits the individual
Health questionnaire (Eq5D-5L) | 2 years
  The EQ-5D is a standardized instrument that scores on five health levels (mobility, self-care, daily activities, pain/discomfort, and anxiety/depression). From this, a weighted health index can be derived for an individual or population.
MS Self-Efficacy Scale (MSSES) | 2 years
  Confidence in being able to undertake daily activities and have control over activities related to MS.
Medical Consumption Questionnaire (iMCQ) | 2 years
  The iMCQ is a non-disease-specific questionnaire that aims to estimate the direct costs of medical care.
Productivity Costs Questionnaire (iPCQ) | 2 years
  The iPCQ aims to measure and subsequently value the indirect costs outside of healthcare: productivity costs
Patient satisfaction questionnaire (PTO) | 2 years
  Patient satisfaction questionnaire about care provided

CONTACTS AND LOCATIONS:
Overall Officials: Dr E. (Esther) Zeinstra, Study Director — Isala; Prof. S (Silvia) Evers, Study Director — Maastricht
Locations (4):
- Netherlands (4):
  - University Medical Center Groningen, Groningen, Nederland
  - University of Maastricht, Maastricht, Nederland
  - MS4research Institute, Nijmegen, Nederland
  - Isala, Zwolle, Nederland

REFERENCES:
- [Derived] Hoving M, Jongen PJ, Evers SMAA, Edens MA, Zeinstra EMPE. MSmonitor-plus program and video calling care (MPVC) for multidisciplinary care and self-management in multiple sclerosis: study protocol of a single-center randomized, parallel-group, open label, non-inferiority trial. BMC Neurol. 2022 Nov 12;22(1):423. doi: 10.1186/s12883-022-02948-z. PMID 36371162